CLINICAL TRIAL: NCT01289483
Title: Fospropofol for Sedation During Elective Awake Intubation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor has decided not to support this study.
Sponsor: The Cleveland Clinic (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10-808
Record Dates: First submitted 2011-01-31; First posted 2011-02-03 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Impaired Airway Clearance
Keywords: awake fiberoptic intubation (AFI); difficult airway; fospropofol
MeSH Terms: interventions — fospropofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- fospropofol 6.5 mg/kg. (Active Comparator): Patient randomized to receive fospropofol for awake intubation at 6.5 mg/kg.
  Interventions: Drug: fospropofol
- fospropofol 5 mg/kg. (Active Comparator): Patient randomized to receive fospropofol for awake intubation at 5 mg/kg.
  Interventions: Drug: fospropofol
- fospropofol 3.5 mg/kg. (Active Comparator): Patient randomized to receive fospropofol for awake intubation at 3 mg/kg.
  Interventions: Drug: fospropofol
- fospropofol 2 mg/kg. (Active Comparator): Patient randomized to receive fospropofol for awake intubation at 2 mg/kg.
  Interventions: Drug: fospropofol

INTERVENTIONS:
Drug: fospropofol — After the initial bolus dose of study drug is given, a maximum of two supplemental doses of fospropofol at 25% of the initial dose will be permitted. Fospropofol supplements will be administered every 4 min
  Arms: fospropofol 6.5 mg/kg.
Drug: fospropofol — After the initial bolus dose of study drug is given, a maximum of two supplemental doses of fospropofol at 25% of the initial dose will be permitted. Fospropofol supplements will be administered every 4 min
  Arms: fospropofol 5 mg/kg.
Drug: fospropofol — After the initial bolus dose of study drug is given, a maximum of two supplemental doses of fospropofol at 25% of the initial dose will be permitted. Fospropofol supplements will be administered every 4 min
  Arms: fospropofol 3.5 mg/kg.
Drug: fospropofol — After the initial bolus dose of study drug is given, a maximum of two supplemental doses of fospropofol at 25% of the initial dose will be permitted. Fospropofol supplements will be administered every 4 min
  Arms: fospropofol 2 mg/kg.

SUMMARY:
Patients scheduled for awake fiberoptic intubation (AFI) because of potential difficult airway will be consented prior to intubation ASA Physical Status classification and history of difficult intubation will be recorded at screening. The investigators will also record the results of airway examination including Mallampati classification, thyromental distance, mouth opening, neck circumference, neck range of motion, presence or absence of beard and overbite, history of neck radiation, and mandibular protrusion test Informed consent will be obtained prior to the procedure from those patients who meet the inclusion and exclusion criteria.

Standard hemodynamic monitoring will be used in all patients including EKG, blood pressure, heart rate, respiratory rate and oxygen saturation. Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scale will be used to assess the level of alertness/sedation. Two consecutive MOAA/S scores of 4 will be considered as the desired effect of moderate sedation.

For AFI procedure, IV will be started and oxygen will be administered. 4 L of oxygen will be delivered through nasal canula until the completion of the AFI procedure. Patient head will be positioned in the sniffing position, Topical anesthesia would be achieved using the topical administration of 4 percent lidocaine using atomized and MaDgic nebulizer, and 2% xylocaine Jel applied to the surface of Williams airway in a total dose of lidocaine not exceeding 10 mg/kg. Patients will be randomized to one of the four fospropofol treatment arms: 2, 3.5, 5, or 6.5 mg/kg

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18-64 years of age
* ASA physical status 1-3 ( Except patients with severe cardiac and/or pulmonary disease
* Weight 60-90 Kg
* Elective surgery requiring awake FOI
* Male or female, female patients should not be pregnant (documented by morning of surgery urine pregnancy test result as per routine hospital policy) or lactating

Exclusion Criteria:

* Previous exposure to any experimental drug within 30 days prior to study drug administration
* Raised intracranial pressure
* Patients for whom propofol is contraindicated
* Allergy to midazolam and/or fentanyl

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Rescue intubation needed | every 4 minutes during procedure, day 1
  Requiring rescue midazolam and or fentanyl to facilitate intubation
Hypotension | every 2 minutes, during procedure, day 1
  Development of hypotension ( defined as blood pressure drop of more than >30 % of base line) and/or hypoxemia ( SaO2 < 90% or a drop of >5% of baseline , whichever is lower)

SECONDARY OUTCOMES:
hypertension | every 2 minutes, during procedure day 1
  Development of hypertension ( increase in blood pressure of > 30% of baseline), and/or tachycardia (120 beat/min or increase in heart rate of > 30% of base line, whichever is higher )
Total dose of midazolam and fentanyl used | end of procedure, day 1
  Total dose of midazolam and fentanyl used
ease of intubation | seconds, after intubation, day 1
  anesthesiologists' assessment of ease of intubation on a visual analog scale (VAS) of 0-10, with 0 being very easy, and 10 being very difficult.
Patient recall and satisfaction | end of procedure,day 1
  Patient recall and satisfaction
Time to intubate | seconds, during procedure, day 1
  Time to intubation ( first fospropofol bolus to positive EtCO2 )
Failed intubation | seconds, day 1
  Failed intubation
unresponsiveness | seconds, during procedure, day 1
  Patient becoming un-responsive and /or requiring bag-mask Ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Basem Abdelmalak, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States